CLINICAL TRIAL: NCT07249255
Title: The Effect of Peripheral Intravenous Catheter Bundle on Catheter Insertion Success, Complication Development, and Procedure-Related Pain in Patients Presenting to the Pediatric Emergency Department
Brief Title: Peripheral Intravenous Catheter Bundle
Acronym: deu-acil-bd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülçin Özalp Gerçeker (Other)
Responsible Party: Sponsor-Investigator, Gülçin Özalp Gerçeker, Prof., Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: deu-560
Record Dates: First submitted 2025-09-24; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pediatric; Catheter Complications; Catheter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vein Imaging Device and Vialon Catheter Group (Experimental): Using a PIVC bundle,Vein Imaging Device, and Vialon catheters
  Interventions: Device: Vein Imaging Device; Device: Vialon catheters
- Vein Imaging Device and Standard/Teflon Catheter Group (Experimental): Using a PIVC bundle,Vein Imaging Device, and Teflon catheters
  Interventions: Device: Vein Imaging Device
- Vialon Catheter Group (Experimental): Using a PIVC bundle and Vialon catheters
  Interventions: Device: Vialon catheters
- Standard/Teflon Catheter Group (No Intervention): Using a PIVC bundle and Teflon catheters

INTERVENTIONS:
Device: Vein Imaging Device — Vein Imaging Device before PIVC insertion
  Arms: Vein Imaging Device and Standard/Teflon Catheter Group; Vein Imaging Device and Vialon Catheter Group
Device: Vialon catheters — Vialon catheter use for PIVC insertion
  Arms: Vein Imaging Device and Vialon Catheter Group; Vialon Catheter Group

SUMMARY:
The study was designed to investigate the effects of a PIVC Bundle, which includes a vein visualization device and a vial (BD Neoflon™ Pro catheter), on catheter placement success, complications, procedure-related pain, and catheter length of stay in children aged 1-6 years who are scheduled for peripheral intravenous catheter (PIVC) insertion.

DETAILED DESCRIPTION:
The study sample included four groups: (1) vein visualization device (VGC) and Vialon Catheter Group, (2) VGC and Standard/Teflon Catheter Group, (3) Vialon Catheter Group, (4) Standard/Teflon Catheter Group/Control Group. Data were collected using the Socio-Demographic Data Collection Form, the Forced Intravenous Intervention Score, the PIVC Site Follow-up Form, the Infiltration Scale, the Extravasation Scale, the Phlebitis Scale, and the FLACC Pain Diagnosis Scale.

ELIGIBILITY:
Inclusion Criteria:

* must be between 1 and 6 years old.
* must be inserted PIC

Exclusion Criteria:

* must be shock or severe dehydration, unconsciousness.
* had a central catheter.
* must be inserted at the lower extremities.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
PIVC insertion related pain score | FLACC score evaluated 3 minutes after the PIVC insertion
  The FLACC (Face, Legs, Activity, Cry, Consolability) score related to the PIVC insertion. The scale is scored in a range of 0-10, with 0 representing no pain. Assessment of score: 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
PIVC indwelling time | immediately after the PIC intervention
  PIVC stay time

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin ÖZALP GERÇEKER, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No